CLINICAL TRIAL: NCT00652145
Title: Test Treat Strategy to Prevent Ulcerative Colitis Relapse
Brief Title: Dose Escalation and Remission (DEAR)
Acronym: DEAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: James Lewis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Shire (Industry)
Responsible Party: Sponsor-Investigator, James Lewis, Professor of Medicine and Epidemiology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K24DK078228 (NIH); K24DK078228 (NIH)
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Results first posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increase mesalamine dose by 2.4g/day (Experimental): Increase dose of mesalamine by 2.4 gm per day
  Interventions: Drug: mesalamine
- Maintain mesalmine dose (No Intervention): Maintain current mesalamine dose at 2.4 g/day

INTERVENTIONS:
Drug: mesalamine — Increase dose by 2.4gm per day over baseline dose
  Other Names: Lialda
  Arms: Increase mesalamine dose by 2.4g/day

SUMMARY:
The proposed study will test whether increasing Lialda dose can reduce fecal calprotectin (FCP) levels, a marker of intestinal inflammation that is highly predictive of the risk of relapse among patients with quiescent ulcerative colitis. Sixty patients with FCP levels <50µg/g stool will be observed for 48 weeks. All patients will have FCP concentration measured using a commercially available assay at enrollment, 6 weeks and 12 weeks. All patients with persistently elevated FCP will receive one or both of the following interventions: change in the mesalamine formulation to Lialda and/or increase in the dose of Lialda. Reduction in FCP levels below 50µg/g stool 6 weeks after randomization will be the primary outcome. The proportion of patients achieving this outcome will be compared between groups using Fisher's exact test. All randomized patients as well as those who were excluded from the randomized trial because of a low FCP concentration at baseline will be followed to week 48 to determine the rate of clinical relapse.

DETAILED DESCRIPTION:
Among patients with quiescent ulcerative colitis (UC), lower fecal concentrations of calprotectin are associated with lower rates of relapse. We performed an open-label, randomized controlled trial to investigate whether increasing doses of mesalamine reduce concentrations of fecal calprotectin (FC) in patients with quiescent UC.

We screened 119 patients with UC in remission on the basis of Simple Clinical Colitis Activity Index scores, FC >50 µg/g, and intake of no more than 3 g/day mesalamine. Participants taking mesalamine formulations other than multimatrix mesalamine were switched to multimatrix mesalamine (2.4 g/day) for 6 weeks; 52 participants were then randomly assigned (1:1) to a group that continued its current dose of mesalamine (controls, n = 26) or a group that increased its dose by 2.4 g/day for 6 weeks (n = 26). The primary outcome was continued remission with FC <50 µg/g. Secondary outcomes were continued remission with FC <100 µg/g or <200 µg/g (among patients with pre-randomization values above these levels).

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign the informed consent form.
2. Have documented ulcerative colitis on the basis of usual diagnostic criteria including clinical symptoms and findings from endoscopy, radiology studies, and histology.
3. Have a Simple Clinical Colitis Activity Index (SCCAI)55 score below 3 with no category value greater than 1 (Table 5).
4. Three or fewer bowel movements per 24 hours at the time of enrollment.
5. No visible blood in their bowel movements in the three days prior to enrollment.
6. Have either been on a stable dose of mesalamine medication (oral, rectal or a combination of oral and rectal, including sulfasalazine) or on no mesalamine medications for at least 4 weeks prior to enrollment.
7. Have been on either a stable dose of azathioprine, 6-mercaptopurine, or methotrexate or on none of these medications for at least 8 weeks prior to enrollment.
8. Have experienced at least one flare of ulcerative colitis in the 2 years prior to enrollment. A flare is defined as an increase in stool frequency, bleeding, urgency and/or abdominal discomfort sufficient to warrant a change in medication dose or addition of a new medication.
9. Most recently measured serum creatinine level in the preceding year less than 1.5 mg/dL.

Exclusion Criteria:

1. Age less than 18
2. Inability to speak and read English
3. Presence of an ostomy or prior total or subtotal colectomy
4. Current corticosteroid use or use within the two weeks prior to enrollment
5. Remission for less than 4 weeks prior to enrollment
6. Previous intolerance to mesalamine at doses greater than the current dose.
7. Use of rectally administered mesalamine or steroids within the 2 weeks prior to enrollment.
8. Currently taking more than 3.0 gm/day of mesalamine (oral or rectal). If on oral and rectal mesalamine, the combined dose is more than 3.0 gm/day.
9. Use of anti-TNFα therapies within the 8 weeks prior to enrollment and/or intent to use anti-TNFα therapies as maintenance therapy in the coming 12 weeks.
10. Pregnant or breast feeding women.
11. Use of an experimental therapy for ulcerative colitis in the 8 weeks prior to enrollment.
12. Any condition that the investigator feels will make completion of the study unlikely.
13. Use of cyclosporine in the two weeks prior to enrollment.
14. Moderate or severe abdominal tenderness on examination at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2008-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Lewis, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (8):
- United States (8):
  - Gastroenterology Group of Naples, Naples, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Maryland Medical Center, Baltimore, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - South Jersey Gastroenterology, Marlton, New Jersey
  - University of Pennsylvania - Presbyterian Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Osterman MT, Aberra FN, Cross R, Liakos S, McCabe R, Shafran I, Wolf D, Hardi R, Nessel L, Brensinger C, Gilroy E, Lewis JD; DEAR Investigators. Mesalamine dose escalation reduces fecal calprotectin in patients with quiescent ulcerative colitis. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1887-93.e3. doi: 10.1016/j.cgh.2014.03.035. Epub 2014 Apr 30. PMID 24793028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We screened 150 patients and enrolled 119 patients with UC in remission on the basis of SCCAI score. 58 patients had baseline fecal calprotectin(FC) <50 µg/g. These patients were followed in an observational arm. 61 had FC >= 50 µg/g,whose current mesalamine dose <3g/day. See preassignment details.
Pre-assignment Details: Among 61 pts with FC >=50 µg/g at week 0, 26 were taking non-MMX mesalamine at baseline and switched to MMX mesalamine 2.4g/day. Of these, by week 6, 2 had a repeat FC <50 µg/g, 3 had a flare of UC and 4 were noncompliant with study protocol or no longer interested in participating. The remaining 52 patients were included in the randomized trial.
Groups:
- Increase Dose of Mesalamine: Increase dose of mesalamine by 2.4gm per day over baseline dose for six weeks
- Maintain Baseline Mesalamine Dose: Maintain baseline mesalamine dose for six weeks
Period: Overall Study
Arm/Group | Increase Dose of Mesalamine | Maintain Baseline Mesalamine Dose
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Increase Mesalamine Dose: Participants were randomized to increase dose of mesalamine by 2.4 gm per day over their baseline dose
- Maintain Mesalamine Dose: Participants were randomized to maintain their baseline mesalamine dose
- Total: Total of all reporting groups
Arm/Group | Increase Mesalamine Dose | Maintain Mesalamine Dose | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43.8 [30.5 to 57.1] | 48.8 [33.5 to 60.4] | 46.5 [32.0 to 58.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 15 | 13 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 22 | 21 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52
Tobacco use [Number; unit: participants]
  Current | 0 | 2 | 2
  Prior | 6 | 8 | 14
  Never | 20 | 16 | 36
Extent of disease [Number; unit: participants]
  Proctitis | 8 | 2 | 10
  Left-sided | 9 | 12 | 21
  Extensive | 9 | 11 | 20
  Other | 0 | 1 | 1
Median duration of UC [Median (Inter-Quartile Range); unit: years] | 11.9 [3.7 to 19.8] | 6.5 [2.2 to 11.9] | 8.9 [2.8 to 15.9]
Median of duration of remission at baseline [Median (Inter-Quartile Range); unit: years] | 0.3 [0.2 to 1.0] | 0.5 [0.2 to 1.1] | 0.4 [0.2 to 1.0]
Median fecal calprotectin immediately before randomization [Median (Inter-Quartile Range); unit: µg/g] | 174 [67.0 to 439] | 214 [80.0 to 439] | 195 [69 to 461]
Currrent oral mesalamine [Number; unit: participants]
  Non-MMX formulation | 8 | 9 | 17
  MMX formulation | 14 | 12 | 26
  None | 4 | 5 | 9
Current rectal mesalamine [Number; unit: participants]
  Yes | 2 | 2 | 4
  No | 24 | 24 | 48
Current thiopurine [Number; unit: participants]
  Yes | 6 | 4 | 10
  No | 20 | 22 | 42
Prior corticosteroids [Number; unit: participants]
  Yes | 11 | 17 | 28
  No | 15 | 9 | 24
Prior rectal corticosteroids [Number; unit: participants]
  Yes | 6 | 7 | 13
  No | 20 | 19 | 39
Prior cyclosporine [Number; unit: participants]
  Yes | 0 | 1 | 1
  No | 26 | 25 | 51
Prior anti-tumor necrosis factor agent [Number; unit: participants]
  Yes | 2 | 0 | 2
  No | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Fecal Calprotectin Level <50µg/g
Time Frame: 6 weeks after randomization
Measure: Number; unit: participants
Arm/Group | Increase Mesalamine Dose by 2.4g/Day | Maintain Mesalmine Dose
Number analyzed (Participants) | 26 | 26
participants | 7 | 1

2. Secondary Outcome: Fecal Calprotectin Level <100 µg/g
Time Frame: at 6 weeks after randomization
Population: 38 participants with baseline FC>=100ug/g
Measure: Number; unit: participants
Arm/Group | Increase Dose of Mesalamine | Maintain Baseline Mesalamine Dose
Number analyzed (Participants) | 19 | 19
participants | 10 | 3

3. Secondary Outcome: Fecal Calprotectin <200 µg/g
Time Frame: at 6 weeks after randomization
Population: 25 participants with baseline FC>=200ug/g
Measure: Number; unit: participants
Arm/Group | Increase Dose of Mesalamine | Maintain Baseline Mesalamine Dose
Number analyzed (Participants) | 13 | 12
participants | 10 | 2

ADVERSE EVENTS:
Description: Participants were asked at each visit if they experienced any new symptoms or whether they were diagnosed with any new medical conditions since their last visit. At each visit, participants were also asked if they had any of the following conditions over the prior 3 days:
  Erythema nodosum Pyoderma gangrenosum Uveitis IBD-associated arthritis
Arm/Group | Increase Dose of Mesalamine | Maintain Baseline Mesalamine Dose
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 11/26 | 7/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Increase Dose of Mesalamine (N=26) | Maintain Baseline Mesalamine Dose (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
blood in stool (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
dizziness (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
headache (General disorders) | 1 (1) | 0 (0)
iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
itchy eyes (Eye disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vitamin B12 deficiency (General disorders) | 1 (1) | 0 (0)
Worsening Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower back pain (General disorders) | 0 (0) | 1 (1)
increase mucous (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry eyes (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No